CLINICAL TRIAL: NCT02494193
Title: Indirect Pulp Capping With Resin Modified Glass Ionomer: a Randomized Controled Clinical Trial
Brief Title: Indirect Pulp Capping With Resin Modified Glass Ionomer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sergipe (Other)
Responsible Party: Principal Investigator, André Luis Faria e Silva, Dr., Universidade Federal de Sergipe
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPC
Record Dates: First submitted 2015-06-30; First posted 2015-07-10 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Caries, Dental; Pulpitis
MeSH Terms: conditions — Dental Caries; Pulpitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular Treatment (Active Comparator): Partial caries removal; Provisional restoration - control; Total caries removal; Definitive restoration.
  Interventions: Other: Partial caries removal; Other: Provisional restoration - control; Other: Total caries removal; Other: Definitive restoration
- Alternative Treatment (Experimental): Partial caries removal; Provisional restoration - experimental; Total caries removal; Definitive restoration.
  Interventions: Other: Partial caries removal; Other: Provisional restoration - experimental; Other: Total caries removal; Other: Definitive restoration

INTERVENTIONS:
Other: Partial caries removal — The caries infected dentin will be removed mantaining the affected caries tissue.
Other: Provisional restoration - control — After partial caries removal, a provisional restoration will be performed using a layer of calcium hydroxide paste covered by a layer of calcium hydroxide cement and resin-modified glass ionomer.
  Arms: Regular Treatment
Other: Provisional restoration - experimental — After partial caries removal, a provisional restoration will be performed using only resin-modified glass ionomer.
  Arms: Alternative Treatment
Other: Total caries removal — After two months of their placement, the provisional restoration will removed followed by tota caries tissue removal.
Other: Definitive restoration — Definite restoration will be performed using composite.

SUMMARY:
In deep carious lesions, presenting risk of pulp exposition, a treatment option is the partial caries removal of carious tissue followed by provisional restoration, while this approach is called indirect pulp capping. The aim of this double-blinding controlled randomized clinical trial is to evaluate the success of indirect pulp capping using only resin-modified glass ionomer, while the additional layer of calcium hydroxide was used as control. The sample of 112 molars and/or premolars (n=56), presenting deep carious lesions, from patients with age between 15 and 30 years treated in dental clinic at Department of Dentistry of Federal University of Sergipe. The selected carious lesions must be reached 2/3 of dentin, observed in bite-wing radiography, without pulp involving and/or other factor that to compromise the evaluation. After detailed anamneses, the selected teeth will be radiographed e all carious tissue from surrounding walls will be removed. At the floor of cavity, the carious tissue will be partially removed using hand dentin excavators, remaining the caries-affected dentin and avoiding the pulp exposition. The removed carious tissue from the floor of cavity will be evaluated for presence of Lactobacilos e Estreptococos Mutans, while the remaining dentin will be evaluated for consistency, colour and humidity. Randomly, the cavity will be provisionally restored with: Control - dress and cement of calcium hydroxide followed resin-modified glass ionomer; or Experimental - only resin-modified glass ionomer. The distance between the base of restoration and the pulp cavity cap will be measured by bitw-wing radiography. The patients will be re-evaluated after 15 days, while the teeth with compromised pulp vitality will be excluded from the study. The remaining patients will be evaluated after 6 months. The distance between the base of restoration and the pulp cavity cap will be measured again, followed by provisional restoration removal. The remaining caries-affected dentin from floor of cavity will be fully removed and a bacteriological evaluation performed. The consistency, colour and humidity of this tissue will be evaluated too. Finally, the permanent restorations will performed.

ELIGIBILITY:
Inclusion Criteria:

* Molars and pre-molars presenting carious lesions involving 2/3 inner of dentin tissue.

Exclusion Criteria:

* Teeth presenting signs of irreversible pulpits or necrose, cervical lesion and/or root exposition, or with carious lesion reaching the pulp.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 112 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Tooth vitality - analysis for positive or negative response | 2 months after placement of provisional restoration

SECONDARY OUTCOMES:
Consistency of dentin tissue - scores of 1 (softned) to 4 (hard) | Immediately after caries removal
Coloration of dentin tissue - scores of 1 (clear yellow) to 5 (darkd) | Immediately after caries removal
Counting of Streptococcus mutans colonies - number of colony-forming units (CFUs) | Immediately after caries removal
Counting of Lactobacillus spp colonies - number of colony-forming units (CFUs) | Immediately after caries removal

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Sergipe, Aracaju, Sergipe, Brazil